CLINICAL TRIAL: NCT00770263
Title: Phase I Study of Erlotinib and Temsirolimus in Resistant Solid Malignancies
Brief Title: Erlotinib and Temsirolimus for Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-1092 / 201108327
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2014-12

CONDITIONS: Solid Tumors
Keywords: any solid tumors
MeSH Terms: interventions — Erlotinib Hydrochloride; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose Level 1A (Experimental): Erlotinib 100 mg administered orally on a once daily schedule for 35 days for the first cycle.
  Erlotinib 100 mg administered orally on a once daily schedule for 28 days for subsequent cycles.
  Temsirolimus 10 mg IV on days 8, 15, 22, and 29 during the first cycle.
  Temsirolimus 10 mg IV on days 8, 15, and 22 during subsequent cycles.
  Interventions: Drug: Erlotinib; Drug: Temsirolimus
- Dose Level 1 (Experimental): Erlotinib 100 mg administered orally on a once daily schedule for 35 days for the first cycle.
  Erlotinib 100 mg administered orally on a once daily schedule for 28 days for subsequent cycles.
  Temsirolimus 15 mg IV on days 8, 15, 22, and 29 during the first cycle.
  Temsirolimus 15 mg IV on days 8, 15, and 22 during subsequent cycles.
  Interventions: Drug: Erlotinib; Drug: Temsirolimus
- Dose Level 2 (Experimental): Erlotinib 100 mg administered orally on a once daily schedule for 35 days for the first cycle.
  Erlotinib 100 mg administered orally on a once daily schedule for 28 days for subsequent cycles.
  Temsirolimus 20 mg IV on days 8, 15, 22, and 29 during the first cycle.
  Temsirolimus 20 mg IV on days 8, 15, and 22 during subsequent cycles.
  Interventions: Drug: Erlotinib; Drug: Temsirolimus
- Dose Level 3 (Experimental): Erlotinib 100 mg administered orally on a once daily schedule for 35 days for the first cycle.
  Erlotinib 100 mg administered orally on a once daily schedule for 28 days for subsequent cycles.
  Temsirolimus 25 mg IV on days 8, 15, 22, and 29 during the first cycle.
  Temsirolimus 25 mg IV on days 8, 15, and 22 during subsequent cycles.
  Interventions: Drug: Erlotinib; Drug: Temsirolimus
- Dose Expansion Phase (Experimental): Erlotinib 100 mg administered orally on a once daily schedule for 35 days for the first cycle.
  Erlotinib 100 mg administered orally on a once daily schedule for 28 days for subsequent cycles.
  Temsirolimus 25 mg IV on days 8, 15, 22, and 29 during the first cycle.
  Temsirolimus 25 mg IV on days 8, 15, and 22 during subsequent cycles.
  Interventions: Drug: Erlotinib; Drug: Temsirolimus

INTERVENTIONS:
Drug: Erlotinib
  Other Names: Tarceva®
Drug: Temsirolimus
  Other Names: Torisel™

SUMMARY:
Define the maximum tolerated dose and dose limiting side-effects of temsirolimus in combination wtih erlotinib in patients with resistant solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Histologic Diagnosis: Patients must have a histologically or cytologically proven solid malignancy which is resistant to conventional therapy or for which no effective therapy is known.
* Dose Expansion Phase ONLY: Patients must have archived tumor tissue available (paraffin blocks, unstained tissue sections, tissue cores).
* Tumor Mutational Status (Dose Expansion Phase ONLY): Patients must have tumor harboring PTEN loss, PIK3CA mutation, , and/or EGFR mutation. Patients cannot have KRAS or BRAF mutations. Patients must have mutational status determined by Genomic and Pathology Services at Washington University (GPS@WU) or other CLIA-certified laboratories.
* Dose Expansion Phase ONLY: Patients with squamous carcinoma histology, papillary thyroid carcinoma, and adenoid cystic carcinoma are eligible for the expansion cohort regardless of genetic alterations..
* Measurable or Non-Measurable Disease: Patients with measurable or non-measurable disease are eligible for entry to this study. In addition, patients without measurable or non-measurable disease are also eligible.
* Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥20 mm with conventional techniques (PET, CT, MRI, x-ray) or as ≥10 mm with spiral CT scan. All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters).
* Tumor markers may be considered non-measurable disease.
* A positive bone scan, osteoblastic metastases, and pleural or peritoneal effusions are not considered measurable or non-measurable. Patients with only these lesions are eligible for entry to the study.
* Dose Expansion Phase ONLY: Patients must have a tumor that is easily accessible for biopsy determined by the treating physician or the study PI. Patients must agree to a mandatory biopsy at the end of cycle 1 treatment.
* Recovery from Prior Therapy: Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. No chemotherapy or radiotherapy may be given within 3 weeks prior to the start of protocol treatment. No prior therapy with erlotinib or temsirolimus allowed.
* Age: Patients must be ≥18 years old. Because no dosing or toxicity data are currently available on the use of temsirolimus in combination with erlotinib in patients <18 years of age, children are excluded from this study, but will be eligible for the pediatric phase I single-agent trials, when available.
* Performance Status: ECOG 0-1 at study entry.
* Life Expectancy: Patients must have a life expectancy of greater than 12 weeks.
* Required Laboratory Values:
* absolute neutrophil count ≥1,500/mm3
* platelets ≥100,000/mm3
* hemoglobin ≥9.0 g/dL
* total bilirubin ≤1.5 x ULN
* AST/ALT ≤3.0 x ULN
* alkaline phosphatase ≤2.5 x ULN
* creatinine ≤2.0 x ULN OR
* creatinine clearance ≥60 mL/min/1.732 for patients with creatinine levels above 2.0 mg/dl
* serum cholesterol ≤350 mg/dL /9.0 mmol/L (fasting)
* triglycerides ≤300 mg/dL (fasting)*
* PT/INR ≤1.5, unless the patient is on full dose warfarin or stable dose of LMW heparin with a therapeutic INR of >1.5 - ≤3

  *Patients with triglyceride levels >400 mg/dL can be started on lipid lowering agents and reevaluated within 1 week. If levels go to ≤400 mg/dL, they can be considered for the trial and continue the lipid lowering agents.
* Temsirolimus is primarily metabolized by CYP3A4. Patients cannot be receiving enzyme-inducing antiepileptic drugs (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital) nor any other CYP3A4 inducer such as rifampin or St. John's wort, as these may decrease temsirolimus levels. A partial list of agents which interact with cytochrome P450 (CYP3A) is found in Appendix AB. Use of agents that potently inhibit CYP3A (and hence may raise temsirolimus levels), such as ketoconazole, is discouraged, but not specifically prohibited. Temsirolimus can inhibit CYP2D6, and may decrease metabolism (and increase drug levels) of drugs that are substrates for CYP2D6, such as codeine. The appropriateness of use of such agents is left to physician discretion. A list of drugs that may have potential interactions with CYP2D6 is found in Appendix A. If there is any doubt about eligibility based on concomitant medication, the Principal Investigator, Dr. Andrea Wang-Gillam, should be contacted. All concomitant medications must be recorded.
* Known Allergies: Patients with known hypersensitivity reactions to macrolide antibiotics (such as erythromycin, clarithromycin, and azithromycin) are not eligible for this trial.
* Sexually Active Patients: For all sexually active patients, the use of adequate contraception (hormonal or barrier method of birth control) will be required prior to study entry and for the duration of study participation. Non-pregnant status will be determined in all women of childbearing potential. Pregnant and nursing women are not eligible.
* HIV-Positive Patients: Patients receiving anti-retroviral therapy (HAART) for HIV infection are excluded from the study because of possible pharmacokinetic interactions. Appropriate studies will be undertaken in patients receiving HAART therapy, when indicated.
* Neurologic Status: Patients must not have active CNS disease.
* Recovery from Intercurrent Illness: Patients must have recovered from uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Informed Consent: Patients must have signed a Washington University Human Research Protection Office (HRPO) approved informed consent. The patient should not have any serious medical or psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment.
* Inclusion of Women and Minorities: Entry to this study is open to both men and women and to all racial and ethnic subgroups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To define the maximum tolerated dose and dose-limiting toxicities of temsirolimus in combination with erlotinib in patients with resistant solid malignancies. | 3 years for MTD to be determined, DLT occurs in 1st cycle only
To determine the incidence and severity of other toxicities of temsirolimus in combination with erlotinib in patients with resistant solid malignancies. | 30 days after end of treatment

SECONDARY OUTCOMES:
To assess the pharmacodynamic profile of temsirolimus in combination with erlotinib. | Prior to each cycle
To determine any anti-tumor activity and response to the combination of temsirolimus and erlotinib in treatment of patients with resistant solid malignancies. | End of treatment
To evaluate the relation between pS6K1 and p-Akt to clinical response to temsirolimus. | End of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Wang-Gillam, M.D., Ph.D., Principal Investigator — Washington Univerisity School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Vignot S, Faivre S, Aguirre D, Raymond E. mTOR-targeted therapy of cancer with rapamycin derivatives. Ann Oncol. 2005 Apr;16(4):525-37. doi: 10.1093/annonc/mdi113. Epub 2005 Feb 22. PMID 15728109
- [Background] Sabers CJ, Martin MM, Brunn GJ, Williams JM, Dumont FJ, Wiederrecht G, Abraham RT. Isolation of a protein target of the FKBP12-rapamycin complex in mammalian cells. J Biol Chem. 1995 Jan 13;270(2):815-22. doi: 10.1074/jbc.270.2.815. PMID 7822316
- [Background] Lorenz MC, Heitman J. TOR mutations confer rapamycin resistance by preventing interaction with FKBP12-rapamycin. J Biol Chem. 1995 Nov 17;270(46):27531-7. doi: 10.1074/jbc.270.46.27531. PMID 7499212
- [Background] Janus A, Robak T, Smolewski P. The mammalian target of the rapamycin (mTOR) kinase pathway: its role in tumourigenesis and targeted antitumour therapy. Cell Mol Biol Lett. 2005;10(3):479-98. PMID 16217558
- [Background] O'Reilly KE, Rojo F, She QB, Solit D, Mills GB, Smith D, Lane H, Hofmann F, Hicklin DJ, Ludwig DL, Baselga J, Rosen N. mTOR inhibition induces upstream receptor tyrosine kinase signaling and activates Akt. Cancer Res. 2006 Feb 1;66(3):1500-8. doi: 10.1158/0008-5472.CAN-05-2925. PMID 16452206
- [Background] Oldham S, Hafen E. Insulin/IGF and target of rapamycin signaling: a TOR de force in growth control. Trends Cell Biol. 2003 Feb;13(2):79-85. doi: 10.1016/s0962-8924(02)00042-9. PMID 12559758
- [Background] Bianco R, Melisi D, Ciardiello F, Tortora G. Key cancer cell signal transduction pathways as therapeutic targets. Eur J Cancer. 2006 Feb;42(3):290-4. doi: 10.1016/j.ejca.2005.07.034. Epub 2006 Jan 11. PMID 16376541
- [Background] Sansal I, Sellers WR. The biology and clinical relevance of the PTEN tumor suppressor pathway. J Clin Oncol. 2004 Jul 15;22(14):2954-63. doi: 10.1200/JCO.2004.02.141. PMID 15254063
- [Background] DeGraffenried LA, Fulcher L, Friedrichs WE, Grunwald V, Ray RB, Hidalgo M. Reduced PTEN expression in breast cancer cells confers susceptibility to inhibitors of the PI3 kinase/Akt pathway. Ann Oncol. 2004 Oct;15(10):1510-6. doi: 10.1093/annonc/mdh388. PMID 15367412
- [Background] Manning BD, Tee AR, Logsdon MN, Blenis J, Cantley LC. Identification of the tuberous sclerosis complex-2 tumor suppressor gene product tuberin as a target of the phosphoinositide 3-kinase/akt pathway. Mol Cell. 2002 Jul;10(1):151-62. doi: 10.1016/s1097-2765(02)00568-3. PMID 12150915
- [Background] Hidalgo M, Rowinsky EK. The rapamycin-sensitive signal transduction pathway as a target for cancer therapy. Oncogene. 2000 Dec 27;19(56):6680-6. doi: 10.1038/sj.onc.1204091. PMID 11426655
- [Background] Rowinsky EK. Targeting the molecular target of rapamycin (mTOR). Curr Opin Oncol. 2004 Nov;16(6):564-75. doi: 10.1097/01.cco.0000143964.74936.d1. PMID 15627018
- [Background] Blagosklonny MV, Darzynkiewicz Z. Four birds with one stone: RAPA as potential anticancer therapy. Cancer Biol Ther. 2002 Jul-Aug;1(4):359-61. No abstract available. PMID 12432246
- [Background] Gambacorti-Passerini CB, Gunby RH, Piazza R, Galietta A, Rostagno R, Scapozza L. Molecular mechanisms of resistance to imatinib in Philadelphia-chromosome-positive leukaemias. Lancet Oncol. 2003 Feb;4(2):75-85. doi: 10.1016/s1470-2045(03)00979-3. PMID 12573349
- [Background] Dudkin L, Dilling MB, Cheshire PJ, Harwood FC, Hollingshead M, Arbuck SG, Travis R, Sausville EA, Houghton PJ. Biochemical correlates of mTOR inhibition by the rapamycin ester CCI-779 and tumor growth inhibition. Clin Cancer Res. 2001 Jun;7(6):1758-64. PMID 11410517
- [Background] Yu K, Toral-Barza L, Discafani C, Zhang WG, Skotnicki J, Frost P, Gibbons JJ. mTOR, a novel target in breast cancer: the effect of CCI-779, an mTOR inhibitor, in preclinical models of breast cancer. Endocr Relat Cancer. 2001 Sep;8(3):249-58. doi: 10.1677/erc.0.0080249. PMID 11566616
- [Background] Geoerger B, Kerr K, Tang CB, Fung KM, Powell B, Sutton LN, Phillips PC, Janss AJ. Antitumor activity of the rapamycin analog CCI-779 in human primitive neuroectodermal tumor/medulloblastoma models as single agent and in combination chemotherapy. Cancer Res. 2001 Feb 15;61(4):1527-32. PMID 11245461
- [Background] Elit L. CCI-779 Wyeth. Curr Opin Investig Drugs. 2002 Aug;3(8):1249-53. PMID 12211424
- [Background] Teachey DT, Obzut DA, Cooperman J, Fang J, Carroll M, Choi JK, Houghton PJ, Brown VI, Grupp SA. The mTOR inhibitor CCI-779 induces apoptosis and inhibits growth in preclinical models of primary adult human ALL. Blood. 2006 Feb 1;107(3):1149-55. doi: 10.1182/blood-2005-05-1935. Epub 2005 Sep 29. PMID 16195324
- [Background] Peralba JM, DeGraffenried L, Friedrichs W, Fulcher L, Grunwald V, Weiss G, Hidalgo M. Pharmacodynamic Evaluation of CCI-779, an Inhibitor of mTOR, in Cancer Patients. Clin Cancer Res. 2003 Aug 1;9(8):2887-92. PMID 12912932
- [Background] Raymond E, Alexandre J, Faivre S, Vera K, Materman E, Boni J, Leister C, Korth-Bradley J, Hanauske A, Armand JP. Safety and pharmacokinetics of escalated doses of weekly intravenous infusion of CCI-779, a novel mTOR inhibitor, in patients with cancer. J Clin Oncol. 2004 Jun 15;22(12):2336-47. doi: 10.1200/JCO.2004.08.116. Epub 2004 May 10. PMID 15136596
- [Background] Hidalgo, M., Rowinsky, E, Erlichman,C, Drengler, R, Marshall, B, Marks, R, Edwards, T, Boni, J, et al., Phase I and Pharmocologic Study of CCI-779, a Cell Cycle Inhibitor. 11th NCI-EORTC-AACR Symposium on New Drugs in Cancer Therapy., 2000.
- [Background] Raymond, E., Alexandre, J, Depenbrock, H et al., CCI-779, a Rapamycin Analog with Antitumor Activity: A Phase I Study utilizing a Weekly Schedule. Proc Am Soc Clin Oncol, 2000.
- [Background] Huang S, Houghton PJ. Inhibitors of mammalian target of rapamycin as novel antitumor agents: from bench to clinic. Curr Opin Investig Drugs. 2002 Feb;3(2):295-304. PMID 12020063
- [Background] Hidalgo, M., Rowinsky, E, Erlichman,C, et al., CCI-779, a Rapamycin Analog and Multifaceted Inhibitor of Signal Transduction: a Phase I Study. Proc Am Soc Clin Oncol, 2000. 19.
- [Background] Atkins MB, Hidalgo M, Stadler WM, Logan TF, Dutcher JP, Hudes GR, Park Y, Liou SH, Marshall B, Boni JP, Dukart G, Sherman ML. Randomized phase II study of multiple dose levels of CCI-779, a novel mammalian target of rapamycin kinase inhibitor, in patients with advanced refractory renal cell carcinoma. J Clin Oncol. 2004 Mar 1;22(5):909-18. doi: 10.1200/JCO.2004.08.185. PMID 14990647
- [Background] Pandya KJ, Dahlberg S, Hidalgo M, Cohen RB, Lee MW, Schiller JH, Johnson DH; Eastern Cooperative Oncology Group (E1500). A randomized, phase II trial of two dose levels of temsirolimus (CCI-779) in patients with extensive-stage small-cell lung cancer who have responding or stable disease after induction chemotherapy: a trial of the Eastern Cooperative Oncology Group (E1500). J Thorac Oncol. 2007 Nov;2(11):1036-41. doi: 10.1097/JTO.0b013e318155a439. PMID 17975496
- [Background] Witzig TE, Geyer SM, Ghobrial I, Inwards DJ, Fonseca R, Kurtin P, Ansell SM, Luyun R, Flynn PJ, Morton RF, Dakhil SR, Gross H, Kaufmann SH. Phase II trial of single-agent temsirolimus (CCI-779) for relapsed mantle cell lymphoma. J Clin Oncol. 2005 Aug 10;23(23):5347-56. doi: 10.1200/JCO.2005.13.466. Epub 2005 Jun 27. PMID 15983389
- [Background] Oza, A., Elit, L, Biagi, J, Gotlieb, W, Tonkin, K, Tsao, MN, et al., A Phase II Study of Temsirolimus (CCI-779) in Patients with Metastatic and/or Recurrent Endometrial Cancer - NCI-CTG IND.160. Clin Cancer Res, 2005. 11(24): p. 9099s.
- [Background] Chang SM, Wen P, Cloughesy T, Greenberg H, Schiff D, Conrad C, Fink K, Robins HI, De Angelis L, Raizer J, Hess K, Aldape K, Lamborn KR, Kuhn J, Dancey J, Prados MD; North American Brain Tumor Consortium and the National Cancer Institute. Phase II study of CCI-779 in patients with recurrent glioblastoma multiforme. Invest New Drugs. 2005 Aug;23(4):357-61. doi: 10.1007/s10637-005-1444-0. PMID 16012795
- [Background] Margolin K, Longmate J, Baratta T, Synold T, Christensen S, Weber J, Gajewski T, Quirt I, Doroshow JH. CCI-779 in metastatic melanoma: a phase II trial of the California Cancer Consortium. Cancer. 2005 Sep 1;104(5):1045-8. doi: 10.1002/cncr.21265. PMID 16007689
- [Background] Galanis E, Buckner JC, Maurer MJ, Kreisberg JI, Ballman K, Boni J, Peralba JM, Jenkins RB, Dakhil SR, Morton RF, Jaeckle KA, Scheithauer BW, Dancey J, Hidalgo M, Walsh DJ; North Central Cancer Treatment Group. Phase II trial of temsirolimus (CCI-779) in recurrent glioblastoma multiforme: a North Central Cancer Treatment Group Study. J Clin Oncol. 2005 Aug 10;23(23):5294-304. doi: 10.1200/JCO.2005.23.622. Epub 2005 Jul 5. PMID 15998902
- [Background] Chan S, Scheulen ME, Johnston S, Mross K, Cardoso F, Dittrich C, Eiermann W, Hess D, Morant R, Semiglazov V, Borner M, Salzberg M, Ostapenko V, Illiger HJ, Behringer D, Bardy-Bouxin N, Boni J, Kong S, Cincotta M, Moore L. Phase II study of temsirolimus (CCI-779), a novel inhibitor of mTOR, in heavily pretreated patients with locally advanced or metastatic breast cancer. J Clin Oncol. 2005 Aug 10;23(23):5314-22. doi: 10.1200/JCO.2005.66.130. Epub 2005 Jun 13. PMID 15955899
- [Background] Hudes G, Carducci M, Tomczak P, Dutcher J, Figlin R, Kapoor A, Staroslawska E, Sosman J, McDermott D, Bodrogi I, Kovacevic Z, Lesovoy V, Schmidt-Wolf IG, Barbarash O, Gokmen E, O'Toole T, Lustgarten S, Moore L, Motzer RJ; Global ARCC Trial. Temsirolimus, interferon alfa, or both for advanced renal-cell carcinoma. N Engl J Med. 2007 May 31;356(22):2271-81. doi: 10.1056/NEJMoa066838. PMID 17538086
- [Background] Mendelsohn J, Baselga J. Epidermal growth factor receptor targeting in cancer. Semin Oncol. 2006 Aug;33(4):369-85. doi: 10.1053/j.seminoncol.2006.04.003. PMID 16890793
- [Background] Salomon DS, Brandt R, Ciardiello F, Normanno N. Epidermal growth factor-related peptides and their receptors in human malignancies. Crit Rev Oncol Hematol. 1995 Jul;19(3):183-232. doi: 10.1016/1040-8428(94)00144-i. No abstract available. PMID 7612182
- [Background] Fox SB, Smith K, Hollyer J, Greenall M, Hastrich D, Harris AL. The epidermal growth factor receptor as a prognostic marker: results of 370 patients and review of 3009 patients. Breast Cancer Res Treat. 1994 Jan;29(1):41-9. doi: 10.1007/BF00666180. PMID 8018963
- [Background] Fry DW. Inhibition of the epidermal growth factor receptor family of tyrosine kinases as an approach to cancer chemotherapy: progression from reversible to irreversible inhibitors. Pharmacol Ther. 1999 May-Jun;82(2-3):207-18. doi: 10.1016/s0163-7258(98)00050-3. PMID 10454198
- [Background] Neal DE, Mellon K. Epidermal growth factor receptor and bladder cancer: a review. Urol Int. 1992;48(4):365-71. doi: 10.1159/000282357. PMID 1357809
- [Background] Parra HS, Cavina R, Latteri F, Zucali PA, Campagnoli E, Morenghi E, Grimaldi GC, Roncalli M, Santoro A. Analysis of epidermal growth factor receptor expression as a predictive factor for response to gefitinib ('Iressa', ZD1839) in non-small-cell lung cancer. Br J Cancer. 2004 Jul 19;91(2):208-12. doi: 10.1038/sj.bjc.6601923. PMID 15187994
- [Background] Woodburn JR. The epidermal growth factor receptor and its inhibition in cancer therapy. Pharmacol Ther. 1999 May-Jun;82(2-3):241-50. doi: 10.1016/s0163-7258(98)00045-x. PMID 10454201
- [Background] Wosikowski K, Schuurhuis D, Johnson K, Paull KD, Myers TG, Weinstein JN, Bates SE. Identification of epidermal growth factor receptor and c-erbB2 pathway inhibitors by correlation with gene expression patterns. J Natl Cancer Inst. 1997 Oct 15;89(20):1505-15. doi: 10.1093/jnci/89.20.1505. PMID 9337347
- [Background] Meyers MB, Shen WP, Spengler BA, Ciccarone V, O'Brien JP, Donner DB, Furth ME, Biedler JL. Increased epidermal growth factor receptor in multidrug-resistant human neuroblastoma cells. J Cell Biochem. 1988 Oct;38(2):87-97. doi: 10.1002/jcb.240380203. PMID 2464605
- [Background] Giralt J, Eraso A, Armengol M, Rossello J, Majo J, Ares C, Espin E, Benavente S, de Torres I. Epidermal growth factor receptor is a predictor of tumor response in locally advanced rectal cancer patients treated with preoperative radiotherapy. Int J Radiat Oncol Biol Phys. 2002 Dec 1;54(5):1460-5. doi: 10.1016/s0360-3016(02)03752-5. PMID 12459370
- [Background] Brabender J, Danenberg KD, Metzger R, Schneider PM, Park J, Salonga D, Holscher AH, Danenberg PV. Epidermal growth factor receptor and HER2-neu mRNA expression in non-small cell lung cancer Is correlated with survival. Clin Cancer Res. 2001 Jul;7(7):1850-5. PMID 11448895
- [Background] Saif MW. Erlotinib: the first biologic in the management of pancreatic cancer. Expert Opin Pharmacother. 2008 Jun;9(9):1595-607. doi: 10.1517/14656566.9.9.1595. PMID 18518788
- [Background] Hidalgo M, Siu LL, Nemunaitis J, Rizzo J, Hammond LA, Takimoto C, Eckhardt SG, Tolcher A, Britten CD, Denis L, Ferrante K, Von Hoff DD, Silberman S, Rowinsky EK. Phase I and pharmacologic study of OSI-774, an epidermal growth factor receptor tyrosine kinase inhibitor, in patients with advanced solid malignancies. J Clin Oncol. 2001 Jul 1;19(13):3267-79. doi: 10.1200/JCO.2001.19.13.3267. PMID 11432895
- [Background] Perez-Soler R. The role of erlotinib (Tarceva, OSI 774) in the treatment of non-small cell lung cancer. Clin Cancer Res. 2004 Jun 15;10(12 Pt 2):4238s-4240s. doi: 10.1158/1078-0432.CCR-040017. PMID 15217965
- [Background] Miller VA, Hirsch FR, Johnson DH. Systemic therapy of advanced bronchioloalveolar cell carcinoma: challenges and opportunities. J Clin Oncol. 2005 May 10;23(14):3288-93. doi: 10.1200/JCO.2005.19.240. PMID 15886316
- [Background] Soulieres D, Senzer NN, Vokes EE, Hidalgo M, Agarwala SS, Siu LL. Multicenter phase II study of erlotinib, an oral epidermal growth factor receptor tyrosine kinase inhibitor, in patients with recurrent or metastatic squamous cell cancer of the head and neck. J Clin Oncol. 2004 Jan 1;22(1):77-85. doi: 10.1200/JCO.2004.06.075. PMID 14701768
- [Background] Gordon AN, Finkler N, Edwards RP, Garcia AA, Crozier M, Irwin DH, Barrett E. Efficacy and safety of erlotinib HCl, an epidermal growth factor receptor (HER1/EGFR) tyrosine kinase inhibitor, in patients with advanced ovarian carcinoma: results from a phase II multicenter study. Int J Gynecol Cancer. 2005 Sep-Oct;15(5):785-92. doi: 10.1111/j.1525-1438.2005.00137.x. PMID 16174225
- [Background] Prados MD, Lamborn KR, Chang S, Burton E, Butowski N, Malec M, Kapadia A, Rabbitt J, Page MS, Fedoroff A, Xie D, Kelley SK. Phase 1 study of erlotinib HCl alone and combined with temozolomide in patients with stable or recurrent malignant glioma. Neuro Oncol. 2006 Jan;8(1):67-78. doi: 10.1215/S1522851705000451. PMID 16443950
- [Background] Raizer JJ. HER1/EGFR tyrosine kinase inhibitors for the treatment of glioblastoma multiforme. J Neurooncol. 2005 Aug;74(1):77-86. doi: 10.1007/s11060-005-0603-7. PMID 16078112
- [Background] Dragovich T, McCoy S, Fenoglio-Preiser CM, Wang J, Benedetti JK, Baker AF, Hackett CB, Urba SG, Zaner KS, Blanke CD, Abbruzzese JL. Phase II trial of erlotinib in gastroesophageal junction and gastric adenocarcinomas: SWOG 0127. J Clin Oncol. 2006 Oct 20;24(30):4922-7. doi: 10.1200/JCO.2006.07.1316. PMID 17050876
- [Background] Mancuso A, Sternberg CN. New treatments for metastatic kidney cancer. Can J Urol. 2005 Feb;12 Suppl 1:66-70; discussion 105. PMID 15780170
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Herbst RS, Prager D, Hermann R, Fehrenbacher L, Johnson BE, Sandler A, Kris MG, Tran HT, Klein P, Li X, Ramies D, Johnson DH, Miller VA; TRIBUTE Investigator Group. TRIBUTE: a phase III trial of erlotinib hydrochloride (OSI-774) combined with carboplatin and paclitaxel chemotherapy in advanced non-small-cell lung cancer. J Clin Oncol. 2005 Sep 1;23(25):5892-9. doi: 10.1200/JCO.2005.02.840. Epub 2005 Jul 25. PMID 16043829
- [Background] Gatzemeier U. Targeting the HER1/EGFR receptor to improve outcomes in non-small-cell lung cancer. Oncology (Williston Park). 2003 Nov;17(11 Suppl 12):7-10. PMID 14682117
- [Background] Faivre S, Kroemer G, Raymond E. Current development of mTOR inhibitors as anticancer agents. Nat Rev Drug Discov. 2006 Aug;5(8):671-88. doi: 10.1038/nrd2062. PMID 16883305
- [Background] Buck E, Eyzaguirre A, Brown E, Petti F, McCormack S, Haley JD, Iwata KK, Gibson NW, Griffin G. Rapamycin synergizes with the epidermal growth factor receptor inhibitor erlotinib in non-small-cell lung, pancreatic, colon, and breast tumors. Mol Cancer Ther. 2006 Nov;5(11):2676-84. doi: 10.1158/1535-7163.MCT-06-0166. PMID 17121914
- [Background] Boffa DJ, Luan F, Thomas D, Yang H, Sharma VK, Lagman M, Suthanthiran M. Rapamycin inhibits the growth and metastatic progression of non-small cell lung cancer. Clin Cancer Res. 2004 Jan 1;10(1 Pt 1):293-300. doi: 10.1158/1078-0432.ccr-0629-3. PMID 14734482
- [Background] Sun SY, Rosenberg LM, Wang X, Zhou Z, Yue P, Fu H, Khuri FR. Activation of Akt and eIF4E survival pathways by rapamycin-mediated mammalian target of rapamycin inhibition. Cancer Res. 2005 Aug 15;65(16):7052-8. doi: 10.1158/0008-5472.CAN-05-0917. PMID 16103051
- [Background] Jimeno A, Kulesza P, Wheelhouse J, Chan A, Zhang X, Kincaid E, Chen R, Clark DP, Forastiere A, Hidalgo M. Dual EGFR and mTOR targeting in squamous cell carcinoma models, and development of early markers of efficacy. Br J Cancer. 2007 Mar 26;96(6):952-9. doi: 10.1038/sj.bjc.6603656. Epub 2007 Mar 6. PMID 17342092
- [Background] Robins, H.I., Wen, P.Y, Chang, S.M, Kuhn, K, et al., Phase I study of erlotinib and CCI-779 (temsirolimus) for patients, with recurrent malignant gliomas (MG) (NABTC 04-02). J Clin Oncol, 2007. 25(18s): p. 2057.
- [Background] Azzariti A, Porcelli L, Gatti G, Nicolin A, Paradiso A. Synergic antiproliferative and antiangiogenic effects of EGFR and mTor inhibitors on pancreatic cancer cells. Biochem Pharmacol. 2008 Mar 1;75(5):1035-44. doi: 10.1016/j.bcp.2007.11.018. Epub 2007 Dec 3. PMID 18191814
- [Background] Di Nicolantonio F, Arena S, Tabernero J, Grosso S, Molinari F, Macarulla T, Russo M, Cancelliere C, Zecchin D, Mazzucchelli L, Sasazuki T, Shirasawa S, Geuna M, Frattini M, Baselga J, Gallicchio M, Biffo S, Bardelli A. Deregulation of the PI3K and KRAS signaling pathways in human cancer cells determines their response to everolimus. J Clin Invest. 2010 Aug;120(8):2858-66. doi: 10.1172/JCI37539. Epub 2010 Jul 26. PMID 20664172
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Derived] Park H, Williams K, Trikalinos NA, Larson S, Tan B, Waqar S, Suresh R, Morgensztern D, Van Tine BA, Govindan R, Luo J, Lockhart AC, Wang-Gillam A. A phase I trial of temsirolimus and erlotinib in patients with refractory solid tumors. Cancer Chemother Pharmacol. 2021 Mar;87(3):337-347. doi: 10.1007/s00280-020-04183-0. Epub 2020 Nov 6. PMID 33159216
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu